CLINICAL TRIAL: NCT00456651
Title: Sleep Apnea-Hypopnea Syndrome and the Pathogenesis of Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Collaborators: Fundacion Caubet-Cimera Islas Baleares (Other); Fondo de Investigacion Sanitaria (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IB570/05
Record Dates: First submitted 2007-04-04; First posted 2007-04-05 (Estimated); Last update posted 2007-04-05 (Estimated); Status verified 2007-04

CONDITIONS: Sleep Apnea; Obesity
Keywords: Sleep Apnea; Obesity; Neuropeptides; Hormones
MeSH Terms: conditions — Sleep Apnea Syndromes; Obesity | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: CPAP (Continuous Positive Airway Pressure)

SUMMARY:
The hypothesis of the study is the following: Patients with sleep apnea-hypopnea syndrome have different pattern in the secretion of hormones.

The chronic sleep disorganization that suffer patients with sleep apnea-hypopnea syndrome (SAHS) may affect the central mechanisms that regulate nutritive behavior and energetic balance, causing an alteration in the secretion of hormones that favour the appearance and/or development of obesity.

DETAILED DESCRIPTION:
OBJECTIVES: To compare the plasmatic profiles of different hormones and neuropeptides, related with weight control, metabolism and intake in patients with SAHS as well as in selected control subjects according to weight.

DESIGN: Multicenter, prospective and controlled study. 40 patients with SAHS will be included as well as 40 control subjects.

METHODS: To all subjects included in the study, the following procedures will be performed:

1. Medical History;
2. Anthropometric variables (height, weight, Body Mass Index;
3. Somnolence evaluation using the Epworth scale;
4. Conventional Polysomnography (PSG);
5. Determination every four hours during a 24 hours period of the levels of leptin adiponectin, resistin, insulin, PCR, etc.
6. Conventional biologic evaluation;
7. Patients will be re-evaluated after three months of treatment with CPAP.

ELIGIBILITY:
Inclusion Criteria:

* Apnea-Hypopnea Index > 15
* Body Mass Index < 27 or > 30 Kg/m2

Exclusion Criteria:

* Presence of any chronic disease
* Drug addiction and/or alcoholism
* Refusal to sign informed consent

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2007-02

PRIMARY OUTCOMES:
OBJECTIVES: To compare the plasmatic profiles of different hormones
and neuropeptides, related with weight control, metabolism and intake
in patients with SAHS as well as in selected control subjects according
to weight.

SECONDARY OUTCOMES:
CPAP (Continuous Positive Airway Pressure) effect on studied variables

CONTACTS AND LOCATIONS:
Overall Officials: Mónica de la Peña, MD, Principal Investigator — Hospital Universitario Son Dureta
Locations (1):
- Hospital Universitario Son Dureta, Palma de Mallorca, Balearic Islands, Spain